CLINICAL TRIAL: NCT06538142
Title: Assessment of Photobiomodulation Combined With New Restorative Material for Teeth With Molar Incisor Hypomineralization on Control of Hypersensitivity and Longevity of Restorations: Randomized Controlled Blind Clinical Trial
Brief Title: Photobiomodulation and New Restorative Material for Teeth With MIH on Control of Hypersensitivity and Longevity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NewRestorativeMaterial
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Hypomineralization Molar Incisor; Hypersensitivity Dentin
MeSH Terms: conditions — Molar Hypomineralization; Dentin Sensitivity | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinical assessments after 48 horas as well as four, eight and twelve months after treatment (follow-up) will be performed by an examiner blinded to allocation (single-blind study).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Photobiomodulation + Restoration with self-cure composite resin (Experimental): The participants will receive photobiomodulation + self-cure composite resin restoration.
  Interventions: Procedure: Photobiomodulation + Restoration with Self-cure Composite Resin
- Restoration with Self-cure Composite Resin (Experimental): The participants will receive self-cure composite resin restoration.
  Interventions: Procedure: Restoration with Self-cure Composite Resin
- Photobiomodulation + Restoration with Photopolymerizable Bulk-fill Composite Resin (Experimental): The participants will receive photobiomodulation + restoration in bulk-fill photopolymerizable composite resin restoration.
  Interventions: Procedure: Photobiomodulation + Restoration with Photopolymerizable Bulk-fill Composite Resin

INTERVENTIONS:
Procedure: Photobiomodulation + Restoration with Self-cure Composite Resin — 1. Initial periapical radiograph;
  2. Hypersensitivity reading (visual analogue scale for subjective pain of volunteer and SCASS for examiner's assessment);
  3. Application of photobiomodulation;
  4. Relative isolation (lip bumper, cotton roll and aspirator);
  5. Selective removal of carious tissue with curette (only Code 6 of MIH-SSS criteria);
  6. Cleaning with cotton and water;
  7. Application of primer (Stela; SDI, Melbourne, Vic, Australia) on dentin and/or enamel, wait 5 seconds;
  8. Application of mild compressed air on adhesive for 3 seconds;
  9. Restoration with self-cure composite resin (Stela; SDI, Melbourne, Vic, Australia) extending to adjacent demarcated opacities;
  10. Clinical follow up after 48 hours and at four-month intervals for a period of 12 months;
  11. Hypersensitivity reading after 48 hours and at four-month intervals for a period of 12 months.
  Arms: Photobiomodulation + Restoration with self-cure composite resin
Procedure: Restoration with Self-cure Composite Resin — 1. Initial periapical radiograph;
  2. Hypersensitivity reading (visual analogue scale for subjective pain of volunteer and SCASS for examiner's assessment);
  3. Relative isolation (lip bumper, cotton roll and aspirator);
  4. Selective removal of carious tissue with curette (only Code 6 of MIH-SSS criteria);
  5. Cleaning with cotton and water;
  6. Application of primer (Stela; SDI, Melbourne, Vic, Australia) on dentin and/or enamel, wait 5 seconds;
  7. Application of mild compressed air on adhesive for 3 seconds;
  8. Restoration with self-cure composite resin (Stela; SDI, Melbourne, Vic, Australia) extending to adjacent demarcated opacities;
  9. Clinical follow up after 48 hours and at four-month intervals for a period of 12 months;
  10. Hypersensitivity reading after 48 hours and at four-month intervals for a period of 12 months.
  Arms: Restoration with Self-cure Composite Resin
Procedure: Photobiomodulation + Restoration with Photopolymerizable Bulk-fill Composite Resin — 1. Initial periapical radiograph;
  2. Hypersensitivity reading (visual analogue scale for subjective pain of volunteer and SCASS for examiner's assessment;
  3. Relative isolation;
  4. Application of photobiomodulation;
  5. Selective removal of carious tissue with curette (only Code 6 of MIH-SSS criteria);
  6. Selective etching of enamel adjacent to demarcated opacities with 35% phosphoric acid for 20s;
  7. Active application of universal adhesive (Ambar) on dentin and enamel for 20 seconds (repeat procedure);
  8. Application of mild compressed air on adhesive for 5 seconds;
  9. Photoactivation for 10s;
  10. Restoration with Tetric N Ceram bulk-fill composite resin; with increments up to 4 mm, extending to demarcated opacities;
  11. Photoactivation for 10 seconds;
  12. Clinical follow up after 48 hours and at four-month intervals for a period of 12 months;
  13. Hypersensitivity reading after 48 hours and at four-month intervals for a period of 12 months.
  Arms: Photobiomodulation + Restoration with Photopolymerizable Bulk-fill Composite Resin

SUMMARY:
Introduction: Molar incisor hypomineralization (MIH) is a qualitative defect of enamel development that occurs in the mineralization phase. MIH affects one or more permanent molars and, occasionally, permanent incisors.

Objective: The aim of the proposed study is to determine whether photobiomodulation combined with a new self-cure resin improves hypersensitivity in molars with MIH and caries (primary outcome). Secondary outcomes include assessing the clinical performance of the self-cure composite resin in terms of restoration longevity and comparing the effectiveness of three interventions-photobiomodulation combined with self-cure resin, self-cure resin alone, and photobiomodulation combined with bulkfill photopolymerizable resin-in controlling hypersensitivity over time.

Methods and analysis: Permanent molars with MIH in patients eight to 12 years of age will be allocated to three groups. Group 1: photobiomodulation + self-cure composite resin restoration; Group 2: self-cure composite resin restoration; Group 3: photobiomodulation + restoration in bulk-fill photopolymerizable composite resin. Photobiomodulation will be performed in a single session involving low-level laser administered to four different points. The laser will be used at a wavelength of 808 nm, power of 100 mW and energy of 1 J per points; irradiance will be 3571 mW/cm², with a total radiant exposure of 35.7 J/cm². Data normality will be checked using the Shapiro-Wilk test, and variance homogeneity will be assessed with the Levene test. Descriptive statistics will be used to present the data, with continuous variables expressed as mean and standard deviation, and categorical variables by relative frequency. To compare the VAS and SCASS scales, repeated measures ANOVA will be employed, considering the 3 groups and 5 time points. Bonferroni adjustment will be applied for post-hoc comparisons. Sphericity will be tested with Mauchly's test, and if violated, Greenhouse-Geisser correction will be applied. A significance level of 0.05 will be adopted. Ethics and dissemination: This protocol received approval from the Human Research Ethics Committee of Nove de Julho University (certificate number: xxxxxxx). The legal guardians of the children will agree to participation by signing a statement of informed consent. The results will be published in a peer-review journal and the data will be made available upon request.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children;
* Eight to 12 years of age;
* At least one permanent first molar with MIH (codes 5 and 6 of molar-incisor hypomineralization severity scoring system [MIH-SSS])
* Presence of hypersensitivity
* Direct viewing and access.

Exclusion Criteria:

* Clinically: signs or symptoms of pulp involvement;
* Radiographically: evidence of pulp involvement (initial periapical radiograph);
* Teeth with MIH with no indication for direct restorative treatment (multiple surfaces associated with large extensions);
* Partially erupted teeth;
* Previous restorative treatment.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Hypersensitivity Assessment | Prior to the procedure, 48 hours after restorative treatment and at four-month intervals for the 12-month follow-up period.
  The Visual Analogue Scale (VAS) will be used for the subjective assessment of hypersensitivity on the part of the volunteer and the Schiff Cold Air Sensitivity Scale (SCASS) will be used for the assessment of the operator and examiner. Following isolation of the neighboring teeth with gauze, compressed air will be applied to the tooth with MIH for three seconds. The SCASS is scored as follows: 0 (no reaction); 1 (no reaction, but patient reports discomfort); 2 (patient reacts and moves away from stimulus); and 3 (patient reacts and asks operator to stop).

SECONDARY OUTCOMES:
Clinical Assessment | Clinical follow up after 48 hours and at four-month intervals for a period of 12 months
  The criteria will be the retention of the restorative material in the cavity, rupture of the enamel adjacent to the restoration and the occurrence of secondary caries. The criteria of the modified USPHS index will be used for the assessment. The restoration will be characterized as a failure and the tooth will be excluded from the study if the C score is determined for any of the USPHS criteria. Photographs of the restorations will be taken using a digital single-lens reflex (DSLR) camera (Canon EOS 700D; Canon, Tokyo, Honshu, Japan) to complement the clinical data. The visual demonstration will contribute to any necessary clarifications and make the discussion and documentation of the cases more efficient.

REFERENCES:
- [Derived] Ribeiro CDPV, Mandetta ARH, Pernomiam FC, Camargo CCB, Romano IMF, Sobral APT, Leal ML, Mesquita-Ferrari RA, Fernandes KPS, Horliana ACRT, Motta LJ, Duran CCG, Bussadori SK. Assessment of photobiomodulation combined with new restorative material for teeth with molar incisor hypomineralization on control of hypersensitivity and longevity of restorations: Protocol for a randomized controlled blind clinical trial. PLoS One. 2025 Aug 13;20(8):e0329641. doi: 10.1371/journal.pone.0329641. eCollection 2025. PMID 40802785